CLINICAL TRIAL: NCT00257153
Title: Thrombus Aspiration Before Standard Primary Angioplasty Improves Myocardial Reperfusion in Acute Myocardial Infarction.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Niguarda Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEAR-MI
Record Dates: First submitted 2005-11-18; First posted 2005-11-22 (Estimated); Last update posted 2006-12-04 (Estimated); Status verified 2005-06

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute myocardial infarction; primary angioplasty; myocardial reperfusion; thrombus aspiration

INTERVENTIONS:
Device: Coronary thrombus aspiration catheter

SUMMARY:
In patients with acute ST-segment elevation myocardial infarction (STEMI), percutaneous coronary intervention (PCI) may cause thrombus dislodgment and impaired microcirculatory reperfusion. This study was designed to test the hypothesis that thrombus aspiration before standard PCI may improve acute myocardial reperfusion, measured by ST-segment resolution (STR) and myocardial blush grade (MBG), compared with standard PCI.

DETAILED DESCRIPTION:
Consecutive STEMI patients, admitted within 12 hours of symptom onset and scheduled for primary PCI are randomly assigned to two treatment strategies: standard PCI including stenting and abciximab (group1) or thrombus aspiration with Pronto™ extraction catheter (Vasc.solutions, Minneapolis) before standard PCI (group2). Patients with cardiogenic shock, previous infarction or thrombolytic therapy are excluded.

ELIGIBILITY:
Inclusion Criteria:

* ST-segment elevation myocardial infarction patients undergoing primary angioplasty within 12 hours from symptom onset.

Exclusion Criteria:

* Cardiogenic shock, previous infarction, previous coronary bypass surgery,bundle branch block or pacemaker induced rythm, controindications to IIb/IIIa inhibitors.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160
Dates: Start 2004-03; Study Completion 2005-09

PRIMARY OUTCOMES:
ST-segment resolution immediately after primary angioplasty
Myocardial Blush grade after angioplasty.

SECONDARY OUTCOMES:
Coronary TIMI flow grade,
distal embolization,
no reflow

CONTACTS AND LOCATIONS:
Overall Officials: Pedro L Silva-Orrego, MD, Principal Investigator — Interventional cardiology laboratory, Cardiology Dpt, Niguarda Hospital; Riccardo Bigi, MD, Study Chair — Cardiology Dpt. of medicine and surgery, University school of medicine, Milan, Italy; Paola Colombo, Study Director — Cardiology Dpt. Niguarda hospital; Silvio Klugmann, MD, Study Chair — cardiology Dpt. Niguarda hospital.
Locations (1):
- Cardiology department, Niguarda hospital, Milan, Italy

REFERENCES:
- [Result] Silva-Orrego P, Colombo P, Bigi R, Gregori D, Delgado A, Salvade P, Oreglia J, Orrico P, de Biase A, Piccalo G, Bossi I, Klugmann S. Thrombus aspiration before primary angioplasty improves myocardial reperfusion in acute myocardial infarction: the DEAR-MI (Dethrombosis to Enhance Acute Reperfusion in Myocardial Infarction) study. J Am Coll Cardiol. 2006 Oct 17;48(8):1552-9. doi: 10.1016/j.jacc.2006.03.068. Epub 2006 Sep 26. PMID 17045887